CLINICAL TRIAL: NCT05340257
Title: An Open Label, Single Arm Study, to Evaluate the Pharmacokinetics and Safety of Augmentin Extra Strength (ES)-600 Suspension in Children Presenting With Community Acquired Pneumonia (CAP) and Acute Bacterial Rhinosinusitis (ABRS) in Brazil
Brief Title: A Pharmacokinetics and Safety Study of Augmentin ES-600 in Children With CAP and ABRS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215335
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Infections, Bacterial
Keywords: Amoxicillin; Clavulanic acid; Community Acquired Pneumonia; Acute Bacterial Rhinosinusitis; Pharmacokinetics; Safety; Clinical response; Augmentin ES
MeSH Terms: conditions — Bacterial Infections; Community-Acquired Pneumonia | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: This is a single arm study
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with CAP and ABRS (Experimental)
  Interventions: Drug: Augmentin ES

INTERVENTIONS:
Drug: Augmentin ES — Amoxicillin and clavulanic acid in fixed dose combination will be administered

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety or tolerability through treatment emergent adverse event (TEAE) and to explore primary and secondary clinical response of treatment with Augmentin ES in pediatric population presenting with CAP and ABRS in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* The participant and/or parent(s)/legal guardian(s) are willing and able to comply with the study protocol.
* In accordance with regional/local laws and regulations,
* a. the parent(s)/legal guardian(s) has given signed informed, dated consent; and the participant has
* b.given written assent, if applicable, to participate in the study (for participants between 7 to 12 years)
* Age: Participant must be aged greater than or equal to (>=) 3 months to 12 years, of either gender.
* Participants who are otherwise healthy and presenting with suspected CAP.
* For participants clinically suspected of CAP, at least 3 of the following 4 criteria are applicable:
* a) History of productive cough and/or shortness of breath.
* b)Fever greater than (>)38.5 degree Celsius (○C) (Axillary temperature)
* c) Tachypnea as defined by Respiratory rate (RR) >= 50 breaths/minute in children up to 11 months RR >= 40 breaths/minute in children from 12 months onwards
* d) Chest X-Ray with shadow or lobar condensation, unilateral or bilateral.

For participants of ABRS:

* The participant and/or parent(s)/legal guardian(s) are willing and able to comply with the study protocol.
* In accordance with regional/local laws and regulations,
* a..The parent(s)/legal guardian(s) has given signed informed, dated consent; and the participant has
* b. given written assent, if applicable, to participate in the study (for participants between 7 to 12 years).
* Age: Participant must be between >=3 months to 12 years of either gender.
* Participants who are otherwise healthy and presenting with suspected ABRS.
* For participants of clinically suspected ABRS, the participants would be eligible if any of the following 2 of the 3 criteria stated below are met:
* a.Children with purulent nasal discharge or daytime productive cough (which may worsen at night) or both persisting for 10 days or more without evidence of improvement.
* b. Fever > 38.3○C (Axillary temperature)
* c. Double sickness defined as initial improvement of symptoms and further worsening/ deterioration after 5 days.

Exclusion Criteria:

* Severe ABRS/CAP requiring hospitalization.
* Currently receiving or has received more than one dose of systemic antibiotic therapy within one week prior to the initiation of the study.
* A serious underlying disease as per clinician's judgment.
* Human immunodeficiency virus (HIV) infection/or any other immunosuppressive condition
* Pre-existing renal insufficiency (for example [e.g.], plasma creatinine > 1.5 times upper limit of normal range for age).
* Pre-existing liver disease(s) and/or hepatic dysfunction.
* Any pre-existing malignancy/any participants undergoing any kind of chemotherapy.
* Evidence of leukopenia and/or thrombocytopenia.
* History of previous hypersensitivity reaction to penicillins, cephalosporins or other Beta-lactam antibiotics.
* History of amoxicillin-clavulanate associated cholestatic jaundice/hepatic dysfunction.
* History of phenylketonuria or a known hypersensitivity to aspartame.
* Received, within 48 hours of study entry, or is scheduled to receive during the study period, any medication which may alter bowel function.
* Received, within 48 hours of study entry, or is scheduled to receive during the study period, any medication which may alter renal function like probenecid.
* Participants who have chronic sinusitis (signs and symptoms lasting greater than 28 days prior to screening visit.
* Significant abnormalities of the sinuses and any complications of ABRS.
* Have concurrent streptococcal pharyngitis or acute otitis media (as the standard doses for both of these conditions is 10 days).
* Any other infection or condition, which necessitates use of a concomitant systemic antimicrobial.
* History of infectious mononucleosis.
* History of pseudomembranous colitis.
* Participants that are on warfarin therapy.
* Receipt of an investigational compound (non-food and drug administration [FDA] and non-Brazil National Health Surveillance Agency [ANVISA] approved) or device within the previous 30 days or five half-lives, whichever is longer, preceding the first dose of study intervention or during the study.
* Participants with symptoms suggestive of active Coronavirus disease 2019 (COVID-19) infection (that is (i.e.), fever, cough, etc.)
* Participants with known COVID-19 positive contacts within the past 14 days.
* Female participants who have attained menarche

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-10-14 (Estimated); Primary Completion 2024-07-08 (Estimated); Study Completion 2024-07-08 (Estimated)

PRIMARY OUTCOMES:
Absorption rate constant (Ka) of amoxicillin and clavulanic acid combination | Up to 10 days
Area under the serum concentration-time curve (AUC) of amoxicillin and clavulanic acid combination | Up to 10 days
Maximum serum concentration (Cmax) of amoxicillin and clavulanic acid combination | Up to 10 days
Clearance (CL) of amoxicillin and clavulanic acid combination | Up to 10 days
Volume of distribution (Vd) of amoxicillin and clavulanic acid combination | Up to 10 days
Terminal half-life (t1/2) of amoxicillin and clavulanic acid combination | Up to 10 days

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAE) | Up to Day 14
Number of participants achieving Primary Clinical Response | Day 11 to Day 14
Number of participants achieving Secondary Clinical response | Day 22 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Brazil (2):
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.